CLINICAL TRIAL: NCT04913714
Title: 10+10+30 Infant Vaccines Communication Via Radio in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: Jimma University (Other); Texas A&M University (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OPP1191306
Record Dates: First submitted 2021-05-26; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Infant ALL

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analyst did not know which group received the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): A district where the radio intervention will be broadcast.
  Interventions: Behavioral: 3-month radio intervention on infant vaccination
- Control (No Intervention): A district where the radio intervention will not be broadcast.

INTERVENTIONS:
Behavioral: 3-month radio intervention on infant vaccination — Radio intervention comprising 10-minute drama, 10-minute discussion of the drama by trained health extension workers and 30-minute phone-in from listeners
  Arms: Intervention

SUMMARY:
A cohort study to investigate the effectiveness of radio intervention comprising 10-minute of drama, 10-minute of discussion led by community extension workers, and 30-minute phone-in from listeners on childhood vaccination coverage and timeliness

DETAILED DESCRIPTION:
The evaluation is conducted in 2 districts located in the Oromia region of Ethiopia. One of the districts will be allocated to receive the 3-month radio intervention while the other district that will not have access to the radio intervention will serve as the control.

Data collection includes survey of mothers at two "key" times: at baseline (when infants are at most 5 weeks old; but before beginning the intervention) and at endline (including examination of infant vaccination records) at most 21 days after the end of the radio intervention. The same mothers and infants to be followed at endline.

ELIGIBILITY:
Inclusion Criteria:

Mother, with infant of at most 5 weeks old; Lives in the study district; Consents to participate in study

Exclusion Criteria:

Mother, with infant of more than 5 weeks old; Does not live in study district; Does not consent to participate in study

Ages: 1 Day to 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1320 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Penta 3 vaccine coverage of infant | up to 3 weeks after the intervention ends
  Infant's vaccination record or mother's recall based on interviewer-administered questionnaire

SECONDARY OUTCOMES:
Timeliness of infant vaccines | up to 3 weeks after the intervention ends
  Infant's vaccination record or mother's recall based on interviewer-administered questionnaire
Full coverage of infant vaccines | up to 3 weeks after the intervention ends
  Infant's vaccination record or mother's recall based on a questionnaire
Perceived barriers to vaccination | Immediately before intervention starts, and up to 3 weeks after the intervention ends
  Mother completes interviewer-administered questionnaire at specified times
Perceived susceptibility to vaccine-preventable diseases in children | Immediately before intervention starts, and up to 3 weeks after the intervention ends
  Mother completes interviewer-administered questionnaire at specified times
Perceived benefits of infant vaccines | Immediately before intervention starts, and up to 3 weeks after the intervention ends
  Mother completes interviewer-administered questionnaire at specified times
Perceived severity of vaccine-preventable diseases in children | Immediately before intervention starts, and up to 3 weeks after the intervention ends
  Mother completes interviewer-administered questionnaire at specified times
Cues to action | Immediately before intervention starts, and up to 3 weeks after the intervention ends
  Mother completes interviewer-administered questionnaire at specified times

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Appiah, DrPH, Principal Investigator — Syracuse University
Locations (2):
- Syracuse University, Syracuse, New York, United States
- Jimma University, Jimma, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon reasonable request after data analysis. Email Dr. Bernard Appiah at beappiah@syr.edu
Time Frame: After publication
Access Criteria: Will be accessible as part of open access publishing